CLINICAL TRIAL: NCT02709941
Title: Respiratory Strength Training Mitigates Hypertension and Sleep Fragmentation in Obstructive Sleep Apnea
Brief Title: Inspiratory Muscle Strength Training for Sleep-related Breathing Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, E. Fiona Bailey,PhD, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16GRNT26700007
Record Dates: First submitted 2016-03-02; First posted 2016-03-16 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive Sleep Apnea; Inspiratory Muscle Strength Training; Baroreceptor Sensitivity; Blood Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: the subjects were randomly allocated to either the sham training group or the inspiratory muscle training group using randomization lists for 4 strata (male/female X young/old)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMST Training Group (Active Comparator): Subjects in inspiratory muscle strength training group will complete 30 breaths against a resistance set at 75% of Maximal Inspiratory Pressure (PI Max) everyday for period of 6 weeks.
  Interventions: Other: Inspiratory muscle strength training
- Placebo Training Group (Placebo Comparator): Subjects in placebo training group will complete 30 breaths against a resistance set at 15% of Maximal Inspiratory Pressure (PI Max) everyday for period of 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Inspiratory muscle strength training — Breathing training designed to augment inspiratory muscle strength, and thus targeted muscle groups may benefit from improved force generating capability result in improved breathing.
  Other Names: IMST
  Arms: IMST Training Group
Other: Placebo
  Arms: Placebo Training Group

SUMMARY:
The purpose of the current study is to investigate the effects of a novel breathing training, called inspiratory muscle strength training (IMST), on sleep patterns, breathing and blood pressure for patients diagnosed with mild, moderate and severe sleep apnea.

DETAILED DESCRIPTION:
Aims of the study:

1. To determine the influence of IMST on resting blood pressure and baroreceptor sensitivity.
2. To determine the effect of IMST on sympathetic nervous system by measuring plasma cathecholamines and nerve recording (MSNA).

Population:

30 subjects aged 30-75 years, who have previously been diagnosed with obstructive sleep apnea, as defined by the National Institutes of Health (National Heart Lung, and Blood Institute) will be included in this study.

Study Protocol:

* Pre-training assessment and overnight sleep study
* 5-10 minutes each day breathing training (IMST) at home using a hand-held device for 6 weeks
* Once weekly laboratory visit
* Post-training assessment and overnight sleep study

Pre- and post-training assessment include blood pressure measurement, body weight, neck circumference, cardiorespiratory monitoring, nerve recording, blood draw and sleep surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-75 years
* Diagnosed with Obstructive Sleep Apnea with Apnea Hypopnea Index (AHI) > 15
* Neck circumference > 16 cm

Exclusion Criteria:

* Body mass index (BMI) > 40kg/m2
* Implanted pacemaker
* On anticoagulant medication
* On hypnotic medication
* On immunosuppressive medication
* Acute or recent (3 months prior to study) infection
* History of hypothyroidism
* History of stroke or neuromuscular disease
* Moderate to severe heart failure
* Severe ischemic heart disease
* Severe obstructive and restrictive lung disease
* Cor pulmonale
* Cognitive disorders
* Obstructive nasal disease or history of spontaneous pneumothorax or rib fracture
* History of neurological, respiratory, head /neck, or thoracic surgery

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressures (mmHg) | Weekly blood pressure measures obtained each week for 6 weeks
  Blood pressure measured with blood pressure cuff and syphygmomanometer via standard auscultation technique.

SECONDARY OUTCOMES:
Apnea hypopnea index | Prior to and upon completion of the 6-weeks respiratory strength training.
  Documentation of the total number of apneas and hypopneas experienced by the individuals per hour of sleep and expressed as the apnea-hypopnea index or AHI which has the following ranges; <5 normal; 5-15 mild, 15-30 moderate and >30 severe AHI.
Sleep Quality Survey (PSQI) | Prior to and upon completion of the 6-weeks training.
  This is a rating scale of overall sleep quality ranging from 0-21 with values <5 rated as indicative of normal or good sleep quality and a score of 21 indicative of most severe sleep disturbance.
Plasma cathecholamines (epinephrine, norepinephrine and dopamine) | Blood draw taken prior to and upon completion of the 6-weeks respiratory strength training.
  Plasma catecholamines are determined via morning blood draw taken after 20 minutes supine rest. Reference ranges for plasma catecholamines are as follows: plasma epinephrine is 10-200 pg/ml; plasma norepinephrine 80-250 pg/ml and plasma dopamine 0-20 pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: E. Fiona Bailey, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- Department of Physiology at the University of Arizona, Tucson, Arizona, United States

REFERENCES:
- [Background] Vranish JR, Bailey EF. Daily respiratory training with large intrathoracic pressures, but not large lung volumes, lowers blood pressure in normotensive adults. Respir Physiol Neurobiol. 2015 Sep 15;216:63-9. doi: 10.1016/j.resp.2015.06.002. Epub 2015 Jun 22. PMID 26112283
- [Background] Mello PR, Guerra GM, Borile S, Rondon MU, Alves MJ, Negrao CE, Dal Lago P, Mostarda C, Irigoyen MC, Consolim-Colombo FM. Inspiratory muscle training reduces sympathetic nervous activity and improves inspiratory muscle weakness and quality of life in patients with chronic heart failure: a clinical trial. J Cardiopulm Rehabil Prev. 2012 Sep-Oct;32(5):255-61. doi: 10.1097/HCR.0b013e31825828da. PMID 22785143
- [Background] Parati G, Di Rienzo M, Bonsignore MR, Insalaco G, Marrone O, Castiglioni P, Bonsignore G, Mancia G. Autonomic cardiac regulation in obstructive sleep apnea syndrome: evidence from spontaneous baroreflex analysis during sleep. J Hypertens. 1997 Dec;15(12 Pt 2):1621-6. doi: 10.1097/00004872-199715120-00063. PMID 9488213
- [Derived] Ramos-Barrera GE, DeLucia CM, Bailey EF. Inspiratory muscle strength training lowers blood pressure and sympathetic activity in older adults with OSA: a randomized controlled pilot trial. J Appl Physiol (1985). 2020 Sep 1;129(3):449-458. doi: 10.1152/japplphysiol.00024.2020. Epub 2020 Jul 30. PMID 32730174